CLINICAL TRIAL: NCT01325038
Title: Effects of Increased Muscle Mass on Resting Metabolic Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Fredrik H Nystrom MD PhD, Linköping University, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Beach08
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Subjects
Keywords: resting metabolic rate
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- extra protein supplement (Active Comparator): isometric training with addition of extra protein
  Interventions: Procedure: Isometric exercise
- extra food supplement (Active Comparator): isometric exercise with addition of extra food and calories: one fast food meal/day
  Interventions: Procedure: Isometric exercise

INTERVENTIONS:
Procedure: Isometric exercise — Isometric exercise several times/week for three months

SUMMARY:
Healthy males are randomized to isometric exercise for three months with either extra protein or extra calories in the form of a fast food meal/day in order to study if increase in muscle mass increases resting metabolic rate and if this is affected by presumed increased caloric intake as compared with only proteins.

Body-composition was measured with Dual-Energy X-ray Absorbimetry (DEXA) and RMR was measured by registration of CO2 production and O2 consumption.

ELIGIBILITY:
Inclusion Criteria:

* healthy males

Exclusion Criteria:

* significant disease
* inability to exercise

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
change in resting metabolic rate | 3 months
  measurement of resting metabolic rate at baseline and at the end of the three month trial period

SECONDARY OUTCOMES:
change in muscle mass | 3 months
  measurement of muscle mass with DEXA at baseline and at the end of the three month trial period

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden, Sweden

REFERENCES:
- [Derived] Hambre D, Vergara M, Lood Y, Bachrach-Lindstrom M, Lindstrom T, Nystrom FH. A randomized trial of protein supplementation compared with extra fast food on the effects of resistance training to increase metabolism. Scand J Clin Lab Invest. 2012 Oct;72(6):471-8. doi: 10.3109/00365513.2012.698021. Epub 2012 Aug 30. PMID 22935042